CLINICAL TRIAL: NCT00615849
Title: Phase III Study of Evaluation of the Efficacy of Additional Mechanical Pleurodesis After Thoracoscopic Wedge Resection for the Management of Primary Spontaneous Pneumothorax
Brief Title: Efficacy of the Additional Mechanical Pleurodesis for Surgical Management of Primary Spontaneous Pneumothorax
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sanghoon Jheon, Chief, Department of Thoracic and Cardiovascular Surgery, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KPT
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Primary Spontaneous Pneumothorax
Keywords: pneumothorax, thoracoscopy, pleurodesis
MeSH Terms: conditions — Pneumothorax | interventions — Thoracoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: thoracoscopic surgery — stapled wedge resection of the lung mechanical pleural abrasion

SUMMARY:
For the definite treatment of primary spontaneous pneumothorax(PSP), thoracoscopic bleb obliteration with pleural adhesive procedure is generally accepted as a standard. But additional pleurodesis is potentially useless procedure on the parietal pleura for treating visceral pleural disese. Furthermore, pleural symphysis could deteriorates normal pleural physiology and cause chronic pain. According to our previous study, stapling resection of the bulla without pleurodesis gave comparable result in recurrence comparing with articles with additional pleurodesis. The purpose of this study is to evaluate surgical outcome of thoracoscopic surgery with or without pleural abrasion and to know whether adhesive procedure is essential in the management of PSP.

ELIGIBILITY:
Inclusion Criteria:

* recurrent pneumothorax
* bilateral pneumothorax
* total collapse/tension pneumothorax
* previous history of contralateral pneumothorax
* visible bulla on simple X-ray
* special occupation/situation
* air leakage more than 2 days with drainage catheter for 1st attack patients

Exclusion Criteria:

* patient refusal and reoperation case

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1440 (Actual)
Dates: Start 2006-11; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
recurrence | follow up more than 1 year

SECONDARY OUTCOMES:
complications | follow up more than 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanghoon Jheon, M.D., Ph.D., Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Bundang Hospital, Seungnam, Gyeonggi-do, South Korea